CLINICAL TRIAL: NCT00692185
Title: Atypical Antipsychotic Medication in Anorexia Nervosa
Brief Title: Effectiveness of Olanzapine Versus Placebo in Treating Outpatients With Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Evelyn Attia, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #5116 (MH069868-02); 1R21MH069868-01 (NIH); DSIR A2-AID
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Eating Disorders
Keywords: Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will take olanzapine.
  Interventions: Drug: Olanzapine
- 2 (Placebo Comparator): Participants will take matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — Participants will take 2.5 mg, 5.0 mg, or 10.0 mg of olanzapine once each evening for 8 weeks.
  Other Names: zyprexa
  Arms: 1
Drug: Placebo — Participants will take 2.5 mg, 5.0 mg, or 10.0 mg of placebo once each evening for 8 weeks.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of the antipsychotic medication olanzapine in treating outpatients with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a disease of disordered eating and is characterized by self-starvation, extreme weight loss, and difficulty maintaining a normal weight. Symptoms and behaviors of AN may include distorted body image, obsessive exercise, lack of menstruation among women, binge and purge eating behaviors, and intense fear of weight gain. Furthermore, people with AN are at a high risk of other mental disorders, such as depression and anxiety, and medical complications, such as organ damage, heart failure, and osteoporosis. Current treatments for AN include nutrition counseling, psychotherapy, and medication. Although weight restoration is a treatment priority, no particular therapeutic approach for patients with AN has clear empirical support. Previous studies have suggested that certain medications usually used to treat schizophrenia, also known as atypical antipsychotic drugs, may be helpful in increasing appetite and reducing anxiety related to weight gain and eating in people with AN. Specifically, the atypical antipsychotic medication olanzapine may be effective in improving overall symptoms of AN and in restoring weight to normal levels. This study will compare the effectiveness of the antipsychotic medication olanzapine versus placebo in treating outpatients with AN.

Participation in this study will last 8 weeks. All participants will first undergo baseline assessments that will include questionnaires and interviews about AN symptoms, a physical exam, vital sign measurements, an electrocardiograph (EKG), and a blood draw. Participants will then be assigned randomly to 8 weeks of daily treatment with olanzapine or placebo. Participants will meet with a study doctor weekly over the 8 weeks of treatment. During these visits, the study doctor will monitor participants' progress, medication dosage, vital signs, and side effects. Participants will also fill out weekly questionnaires about the status of their condition and monthly repeat baseline questionnaires. In addition, participants will undergo blood draws every 2 weeks for the first month of the study and every 4 weeks for the remainder of the study. Upon completing the 8 weeks of treatment, participants will repeat the baseline assessments. During the next 5 years, participants may be contacted to complete a follow-up interview.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria (not including amenorrhea) for AN
* Body mass index (BMI) less than 19 kg/m2 and greater than 14 kg/m2
* Patient (or family if the patient is a minor) refuses hospitalization
* Free of psychotropic medication (4 weeks medication free for fluoxetine and antipsychotic medication; 2 weeks medication free for all others) OR on a stable dose of an SSRI or SNRI (venlafaxine) for 4 weeks before study entry
* Prior treatment of AN

Exclusion Criteria:

* Any medical or psychiatric problem requiring urgent attention and/or any significant comorbid illness not likely to benefit from proposed treatments
* Allergy to olanzapine
* Significant orthostatic high blood pressure
* Recent commencement of psychotherapy in the community
* Diabetes mellitus, with a fasting serum glucose greater than 120 mg/dL or nonfasting serum glucose greater than 140 mg/dL
* Known history of current or past jaundice
* Known history of narrow angle glaucoma
* Active substance abuse or dependence
* Schizophrenia, schizophreniform disorder, or bipolar illness
* Movement disorder or presence of tics
* History of tardive dyskinesia
* History of seizures
* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Attia, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (1):
- Eating Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Attia E, Kaplan AS, Walsh BT, Gershkovich M, Yilmaz Z, Musante D, Wang Y. Olanzapine versus placebo for out-patients with anorexia nervosa. Psychol Med. 2011 Oct;41(10):2177-82. doi: 10.1017/S0033291711000390. Epub 2011 Mar 22. PMID 21426603

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine: Dosing of olanzapine began at 2.5 mg daily and was increased every two weeks, first to 5 mg, then 10 mg if the patient was tolerating the medication. If side effects were significant, dosage of the study medication could be lowered. All subjects received 8 weeks of assigned medication.
- Placebo: Participants will take matched placebo for 8 weeks.
Period: Overall Study
Arm/Group | Olanzapine | Placebo
Started | 11 | 12
Completed | 8 | 9
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (9.9) | 26.9 (8.7) | 27.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
  Canada | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain
Time Frame: Measured at Week 8
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Placebo: Participants will take matched placebo for 8 weeks.Dosing of placebo began at 2.5 mg daily and was increased every two weeks, first to 5 mg, then 10 mg . All subjects received 8 weeks of assigned medication.
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 11 | 12
lbs | 6.2 (6.6) | 1.5 (4.4)

2. Secondary Outcome: Symptom Severity Assessed by Yale Brown Cornell-Eating Disorders Scale
Description: The Yale Brown Cornell-Eating Disorders Scale was used.This scale assesses severity of preoccupations and rituals. There are 8 questions that can be scored between 0-4 to indicate severity of symptoms, with 0 representing less severe and 4 representing most severe symptoms. The scores were summed, with possible results totaling 0-32.
Time Frame: Measured at Week 8
Population: Individuals with anorexia nervosa
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Olanzapine: Participants will take olanzapine.
  Dosing of olanzapine began at 2.5 mg daily and was increased every two weeks, first to 5 mg, then 10 mg if the patient was tolerating the medication. If side effects were significant, dosage of the study medication could be lowered. All subjects received 8 weeks of assigned medication
- Placebo: Participants will take matched placebo.
  Placebo: Participants will take 2.5 mg, 5.0 mg, or 10.0 mg of placebo once each evening for 8 weeks.
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 8 | 9
score on a scale | 19.4 (8.1) | 18.9 (6.5)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Olanzapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No